CLINICAL TRIAL: NCT01458171
Title: A Multicenter Follow-up Study of Long-term Safety, Tolerability, and Efficacy of Immune Globulin Subcutaneous (Human) IgPro20 in Subjects With Primary Immunodeficiency
Brief Title: Follow-up Study of Subcutaneous Immune Globulin in Patients Requiring IgG Replacement Therapy (Japan Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLB07_001CR
Record Dates: First submitted 2011-10-12; First posted 2011-10-24 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-02

CONDITIONS: Primary Immune Deficiency Disorder
Keywords: Immune globulin subcutaneous; SCIG; Primary immunodeficiency; PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Hizentra

ARMS (1):
- IgPro20 (Experimental)
  Interventions: Biological: Immune globulin subcutaneous (Human)

INTERVENTIONS:
Biological: Immune globulin subcutaneous (Human) — IgPro20 is a 20% (weight per volume [w/v]) liquid formulation of human immunoglobulin for subcutaneous (SC) use. Subjects will receive weekly infusions of IgPro20 for a total of 24 weeks at a dose based on the subject's IgPro20 dose in the pivotal study ZLB06_002CR (NCT01199705).
  Other Names: Hizentra

SUMMARY:
The objective of this study is to assess the long-term safety, tolerability, and efficacy of IgPro20 in subjects with primary immunodeficiency (PID) as a follow-up to the pivotal study ZLB06_002CR (NCT01199705).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have participated in study ZLB06_002CR and who have tolerated IgPro20 well.
* Written informed consent by the subject/parent/legally acceptable representative. Written assent for an underage subject (≥7 years at the time of obtaining informed consent), as far as possible.

Exclusion Criteria:

* Ongoing serious bacterial infections (SBIs) (pneumonia, bacteremia/septicemia, osteomyelitis/septic arthritis, bacterial meningitis, or visceral abscess) at the time of the first infusion.
* Hypoalbuminemia, protein-losing enteropathies, and any proteinuria (known total urine protein concentration >0.2 g/L or urine protein ++ by dipstick).
* Pregnancy or nursing mother.
* Participation in a study with an investigational medicinal product (IMP) within 3 months prior to enrollment except for ZLB06_002CR.
* Subjects who are planning to donate blood during the study.
* Re-entry of subjects previously participating in the current follow-up study.
* Known or suspected antibodies to the IMP, or to excipients of the IMP.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Midori Kobayashi, Study Director — CSL Behring K.K.
Locations (9):
- Japan (9):
  - Study site, Nagoya, Aichi Pref.
  - Study site, Chiba, Chiba Pref.
  - Study site, Fukuoka, Fukuoka
  - Study site, Gifu, Gifu Pref.
  - Study site, Sapporo, Hokkaido
  - Study site, Moriguchi, Osaka
  - Study site, Koshigaya, Saitama Pref.
  - Study site, Tokorozawa, Saitama Pref.
  - Study site, Bunkyō City, Tokyo Metropolitan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study enrolled subjects at nine study centers in Japan who had participated in the preceding pivotal study ZLB06_002CR (CT.gov identifier: NCT01199705).
Pre-assignment Details: Only subjects participating in the preceding pivotal study ZLB06_002CR (NCT01199705) were eligible. The enrolment visit of this study was on the same day as the completion visit of the preceding pivotal study ZLB06_002CR.
Period: Overall Study
Arm/Group | IgPro20
Started | 23
Completed | 22
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | IgPro20
Number analyzed (Participants) | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 20.8 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Median of the Individual Subject's Rate of Adverse Events (AEs) Per Infusion
Description: The rate was calculated by counting all newly developed or worsened AEs within a subject and dividing by the total number of IgPro20 infusions administered to this subject. Subsequently, the median of these individual AE rates per infusion was calculated. AE rates were classified (i) by severity (mild, moderate, severe) and (ii) by causal relationship to study medication (not related or unlikely related; at least possibly related [i.e., possibly related, probably related, or related]).
Time Frame: 24 weeks
Population: The All Treated (AT) set comprised all subjects receiving at least 1 IgPro20 infusion.
Measure: Median (Full Range); unit: AEs per infusion
Arm/Group | IgPro20
Number analyzed (Participants) | 23
AEs per infusion
  All AEs | 0.167 [0 to 1.71]
  Mild AEs | 0.125 [0 to 1.71]
  Moderate AEs | 0 [0 to 0.04]
  Severe AEs | 0 [0 to 1.00]
  Not related or unlikely related AEs | 0.125 [0 to 0.75]
  At least possibly related AEs | 0 [0 to 1.00]

2. Secondary Outcome: Overall Rate of AEs Per Infusion
Description: The rate was calculated by counting all newly developed or worsened AEs during the treatment period in all subjects and dividing the total number of AEs by the total number of IgPro20 infusions administered. In addition, individual AEs were classified (i) by severity (mild, moderate, severe) and (ii) by causal relationship to study medication (not related or unlikely related; at least possibly related [i.e., possibly related, probably related, or related]). The AE rates per infusion by severity and causal relationship to study medication were calculated by dividing the number of AEs in each category by the total number of IgPro20 infusions.
Time Frame: 24 weeks
Population: The AT set comprised all subjects receiving at least 1 IgPro20 infusion.
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro20
Number analyzed (Participants) | 23
Number analyzed (Infusions) | 529
AEs per infusion
  All AEs | 0.346
  Mild AEs | 0.342
  Moderate AEs | 0.002
  Severe AEs | 0.002
  Not related or unlikely related AEs | 0.210
  At least possibly related AEs | 0.136

3. Secondary Outcome: Number of Subjects With Newly Developing or Worsening AEs
Description: Number of subjects with AEs, overall and classified (i) by severity (mild, moderate, severe) and (ii) by causal relationship to study medication (not related or unlikely related; at least possibly related [i.e., possibly related, probably related, or related]).
Time Frame: 24 weeks
Population: The AT set comprised all subjects receiving at least 1 IgPro20 infusion.
Measure: Number; unit: participants
Arm/Group | IgPro20
Number analyzed (Participants) | 23
participants
  All AEs | 22
  Mild AEs | 21
  Moderate AEs | 1
  Severe AEs | 1
  Not related or unlikely related | 12
  At least possibly related | 10

4. Secondary Outcome: Percentage of Infusions With Subject-assessed Tolerability of at Least 'Good'
Description: Subjects assessed their overall perception of local tolerability at the infusion site throughout the study in the subject diary within a time window of 24 h to 72 h after the end of the latest infusion by assessing it as "very good", "good", "fair", or "poor". The reported percentage represents the percentage of subjects with local tolerability assessments of "very good" or "good" at any given study infusion.
Time Frame: 24 to 72 hours after infusion
Population: The FAS comprised all subjects receiving at least 1 IgPro20 infusion.
Measure: Number; unit: percentage of infusions
Arm/Group | IgPro20
Number analyzed (Participants) | 23
percentage of infusions | 85.4

5. Secondary Outcome: IgG Trough Level
Description: Serum IgG trough levels at the completion visit compared to the baseline visit of the follow-up study. IgG trough levels at baseline, at the completion visit, and the change from baseline to the completion visit are shown
Time Frame: 24 weeks
Population: The Full Analysis Set (FAS) comprised all subjects receiving at least 1 IgPro20 infusion. The Per Protocol Set (PPS) comprised all subjects with the disease under study who a) received uniformly repeated IgPro20 infusions at weekly intervals and b) who had at least 1 documented total serum IgG trough level.
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- IgPro20 - FAS: The FAS comprised all subjects receiving at least 1 IgPro20 infusion.
- IgPro20 - PPS: The PPS comprised all subjects with the disease under study who a) received uniformly repeated IgPro20 infusions at weekly intervals and b) who had at least 1 documented total serum IgG trough level.
Arm/Group | IgPro20 - FAS | IgPro20 - PPS
Number analyzed (Participants) | 23 | 19
g/L
  Baseline | 7.469 (1.3943) | 7.586 (1.3363)
  Completion visit | 8.914 (4.0502) | 8.227 (1.5458)
  Change from baseline to the completion vist | 1.445 (3.4379) | 0.642 (0.7687)

6. Secondary Outcome: Annualized Rate of Clinically Documented Serious Bacterial Infections (SBIs)
Description: SBIs are defined as bacterial pneumonia, bacteremia and septicemia, osteomyelitis/septic arthritis, bacterial meningitis, or visceral abscess. The annualized rate was based on the total number of SBIs and the total number of subject study days for all subjects in the FAS and PPS and adjusted to 365 days.
Time Frame: 24 weeks
Population: The FAS comprised all subjects receiving at least 1 IgPro20 infusion. The PPS comprised all subjects with the disease under study who a) received uniformly repeated IgPro20 infusions at weekly intervals and b) who had at least 1 documented total serum IgG trough level.
Measure: Number; unit: SBIs per subject year
Units Other Than Participants: Total Study Days
Arm/Group | IgPro20 - FAS | IgPro20 - PPS
Number analyzed (Participants) | 23 | 19
Number analyzed (Total Study Days) | 3739 | 3214
SBIs per subject year | 0.00 | 0.00
Statistical Analysis 1: Comparison: IgPro20 - FAS; Test type: Superiority or Other; Annualized Rate = 0.00, 99% CI 1-sided [upper limit 0.450]
Statistical Analysis 2: Comparison: IgPro20 - PPS; Test type: Superiority or Other; Annualized Rate = 0.00, 99% CI 1-sided [upper limit 0.523]

7. Secondary Outcome: Number of Infection Episodes (Serious and Non-serious)
Time Frame: 24 weeks
Population: as for outcome 6
Measure: Number; unit: infection episodes
Arm/Group | IgPro20 - FAS | IgPro20 - PPS
Number analyzed (Participants) | 23 | 19
infection episodes | 43 | 38

8. Secondary Outcome: Number of Days Out of Work/School/Kindergarten/Day Care or Unable to Perform Normal Daily Activities Due to Infections.
Description: Median number of days out of work/school/kindergarten/day care or unable to perform normal daily activities due to infections.
Time Frame: 24 weeks
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | IgPro20 - FAS | IgPro20 - PPS
Number analyzed (Participants) | 23 | 19
days | 0 [0 to 12] | 0 [0 to 9]

9. Secondary Outcome: Number of Days of Hospitalization Due to Infections.
Description: Median number of days of hospitalization due to infections.
Time Frame: 24 weeks
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | IgPro20 - FAS | IgPro20 - PPS
Number analyzed (Participants) | 23 | 19
days | 0 [0 to 11] | 0 [0 to 0]

10. Secondary Outcome: Duration of Use of Antibiotics for Infection Prophylaxis and Treatment
Description: Median number of days of use of antibiotics for infection prophylaxis and/or treatment
Time Frame: 24 weeks
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | IgPro20 - FAS | IgPro20 - PPS
Number analyzed (Participants) | 23 | 19
days | 91.5 [6 to 170] | 154.0 [6 to 170]

11. Other Pre Specified Outcome: Rate of Infection Episodes (Serious and Non-serious)
Description: The annualized rate of infection episodes (serious and non-serious) was based on the total number of infection episodes and the total number of subject study days for all subjects in the FAS population and the PPS population and adjusted to 365 days.
Time Frame: 24 weeks
Population: as for outcome 6
Measure: Number; unit: infection episodes per subject year
Units Other Than Participants: Total Study Days
Arm/Group | IgPro20 - FAS | IgPro20 - PPS
Number analyzed (Participants) | 23 | 19
Number analyzed (Total Study Days) | 3739 | 3214
infection episodes per subject year | 4.20 | 4.32

ADVERSE EVENTS:
Time Frame: For the duration of the study, that is, 24 weeks.
Description: Only AEs starting at or after the first study drug infusion are included. The AT set comprised all subjects receiving at least 1 IgPro20 infusion. AEs in "General disorders" were collected under the MedDRA SOC General disorders and administration site conditions.
Arm/Group | IgPro20
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (N=23)
Encephalitis (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (N=23)
Dental caries (Gastrointestinal disorders) | 4 (4)
Injection site induration (General disorders) | 2 (2)
Injection site pain (General disorders) | 5 (37)
Pyrexia (General disorders) | 2 (4)
Bronchitis (Infections and infestations) | 2 (3)
Conjunctivitis infective (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (13)
Pharyngitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (8)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (8)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.